CLINICAL TRIAL: NCT03456778
Title: Assessing the Efficacy of the Treatment of Tendinopathy With Shear Wave Elastography
Brief Title: Assessing the Tendons With Shear Wave Elastography
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, David Reiter, Associate Professor, Emory University
Other Study IDs: IRB00096405
Record Dates: First submitted 2018-03-02; First posted 2018-03-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Tendinopathy
Keywords: Sonographic imaging; Shear Wave Elastography
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Shear Wave Elastography for Asymptomatic Volunteers: Patients with extremity pain but without tendon involvement will have tendon imagining using shear wave elastography.
  Interventions: Device: Shear Wave Elastography
- Shear Wave Elastography Symptomatic Volunteers: Patients diagnosed with tendinopathy will have tendon imagining using shear wave elastography. Participants may have the option to have repeated imaging to examine tendon healing for up to a year after receiving standard of care treatment.
  Interventions: Device: Shear Wave Elastography

INTERVENTIONS:
Device: Shear Wave Elastography — An ultrasound (US) technique, known as shear wave elastography (SWE), is used to examine structure and biomechanical function. The examination takes place in the ultrasound room at the study site and lasts for approximately 20 minutes.

SUMMARY:
The purpose of this study is to utilize Shear Wave Elastography (SWE) to study the viscoelastic properties of tendons to understand the functional differences between normal/asymptomatic and symptomatic tendon states. The study will also assess the degree of tendon healing following standard of care treatment.

DETAILED DESCRIPTION:
Tendinopathy is a common affliction in athletes, recreational exercisers, the general population and even inactive people. Tendon pathology presenting clinically is most commonly seen in the chronic state related to tendon degeneration manifested as intra-tendinous mucoid degeneration and chondroid metaplasia, which in many cases is accompanied by superimposed small intrasubstance/interstitial tears. Then a vicious cycle of attempted inadequate healing with superimposed acute pathology ensues leading to significant pain and discomfort over time significantly limiting physical activity. The exact pathogenesis of this disease has not been clarified scientifically.

The first part of this study aims to establish the difference between asymptomatic and symptomatic tendons among patients affected by moderate-to-severe, chronic (>6 months of symptoms) tendinopathy in comparison to asymptomatic patients. After establishing a range of elastography normal to severe pathologic measurements, a second part of the study will focus on utilizing ultrasound elastography imaging follow up to assess degree of tendon healing after various standard of care treatments.

The purpose of this prospective observational study is to utilize a ultrasound modality known as real-time Shear Wave Elastography (SWE) to study the viscoelastic properties of tendons, such as the Achilles, patellar, quadriceps, epicondylar, and rotator cuff, to understand the functional differences between normal/asymptomatic (n=75) vs symptomatic (n=75) tendon states (total n=150). The secondary aim will be to assess the degree of tendon healing after standard of care treatment. The clinical implications are very significant because it will provide insights into the mechanism of tendon healing.

ELIGIBILITY:
Inclusion Criteria for Asymptomatic Volunteers:

* Patients presenting at the study location with lower extremity pain without tendon involvement

Inclusion Criteria for Symptomatic Volunteers:

* Patients presenting at the study location with a clinical diagnosis of tenalgia
* Diagnosis of tendinopathy confirmed by ultrasound

Exclusion Criteria:

* Pregnancy
* History of tendinopathy or surgery and morphologic abnormalities
* History of systemic, metabolic, endocrine diseases, or psoriasis
* History of treatment with corticosteroids, estrogens, long term quinolone antibiotics, and cholesterol drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the Emory Orthopaedics and Spine Center who are asymptomatic or symptomatic for tendinopathy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Viscoelastic Tendon Property | Baseline
  Shear wave elastography imaging will be used to establish baseline measurements of viscoelastic properties of tendons, such as the Achilles, patellar, quadriceps, epicondylar, and rotator cuff, among asymptomatic and symptomatic patients.
Change in Tendon Healing | Baseline, Month 3, Month 6, Month 12
  The degree of tendon healing among symptomatic patients receiving standard of care treatment will be assessed by examining stiffness changes measured by shear wave imaging.
Change in Victorian Institute of Sport Assessment - Achilles (VISA-A) Score | Month 6, Month 9, Month 12
  Participants symptomatic for Achilles tendinopathy who received standard of care treatment will be asked to complete the VISA-A scale. The VISA-A scale assesses the severity of chronic Achilles tendinopathy. This 8-item, self-administered questionnaire asks about Achilles tendon pain, daily living function, and sporting activity. Total scores can range from 0 to 100, with 0 representing worst pain and function and 100 signifying no pain or limitations to function. Scores below 70 indicate the presence of Achilles tendinopathy.
Change in Victorian Institute of Sport Assessment - Patellar Tendon (VISA-P) Score | Month 6, Month 9, Month 12
  Participants symptomatic for patellar tendinopathy who received standard of care treatment will be asked to complete the VISA-A scale. The VISA-P scale assesses patellar tendinosis. This 8-item, self-administered questionnaire asks about symptoms, pain, function, and sporting activity. Total scores can range from 0 to 100, with 0 representing worst pain and function and 100 signifying no pain or limitations to function.
Change in The Foot & Ankle Disability Index (FADI) Score | Month 6, Month 9, Month 12
  The FADI is a self-report instrument assessing function related to the foot and ankle. The FADI has 26 items that are scored on a 5-point scale where 0 = unable to do and 4 = no difficulty at all. Total raw scores range from 0 to 104 and scores are converted to percentages, where 100% indicates no dysfunction. This instrument is administered to symptomatic patients receiving standard of care treatment.
Change in The Foot & Ankle Disability Index (FADI) Sport Score | Month 6, Month 9, Month 12
  The FADI Sport is a self-report instrument assessing function related to the foot and ankle in athletes. The FADI Sport has 8 items that are scored on a 5-point scale where 0 = unable to do and 4 = no difficulty at all. Total raw scores range from 0 to 32 and scores are converted to percentages, where 100% indicates no dysfunction. This instrument is administered to symptomatic patients receiving standard of care treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Reiter, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Orthopaedics and Spine Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No